CLINICAL TRIAL: NCT04286880
Title: Comparative Efficacy of Platelet Rich Plasma Injection and Dry Needling in Management of Trigger Points in Masseter Muscle in Myofascial Pain Syndrome Patients
Brief Title: Comparative Efficacy of PRP and Dry Needling in Management of Trigger Points in Masseter Muscle in MPS Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: varsha10av
Record Dates: First submitted 2020-02-18; First posted 2020-02-27 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Myofascial Pain Syndrome
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Dry Needling

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEST GROUP (Experimental): Test group will be administered 0.5 ml of PRP solution per trigger point in masseter muscle.
  Interventions: Procedure: PRP injection
- CONTROL GROUP (Active Comparator): In control group, dry needling will be performed.
  Interventions: Procedure: Dry needling

INTERVENTIONS:
Procedure: PRP injection — Clinically proven cases of Trigger points in masseter muscle will be randomly and equally divided into test group and control group. The selected subjects will be divided into two groups.
  Test group will be administered 0.5 ml of PRP solution per trigger point in masseter muscle according to symptoms of patient at baseline (0 week). PRP will be prepared as per methodology mentioned by Okuda et al 2003.
  Arms: TEST GROUP
Procedure: Dry needling — In control group all the armamentarium and procedure will remain same except that no PRP solution will be delivered. Only dry needling will be performed on the baseline.
  Arms: CONTROL GROUP

SUMMARY:
Title: Comparative Efficacy of Platelet Rich Plasma injection and Dry Needling in management of trigger points in masseter muscle in Myofascial Pain Syndrome patients.

Rationale: Pain and trismus caused by Myofascial pain syndrome in masticatory muscles are one of the prime concerns for the patients. In the recent times, Platelet Rich Plasma therapy has been studied extensively and has produced promising results. It is used to promote sarcomere repair by concentrating growth factors and decrease inflammation by inhibiting pro-inflammatory and apoptotic cells.

Thus, the present study is designed to evaluate the efficacy of Platelet Rich Plasma injection in trigger points in masseter muscle in myofascial pain syndrome patients.

Research Question P: Population (Patients with trigger points in masseter muscle) I: Intervention (PRP injection) C: Control (Dry needling) O: Outcome (Improvement in symptom of pain ) T: Time Frame (1 year) S: Study Design (Randomized clinical trial) Setting in Haryana , India Is Platelet Rich Plasma more effective as compared to dry needling alone in treatment of trigger points in masseter muscle in Myofascial Pain Syndrome patients ?

DETAILED DESCRIPTION:
Myofascial pain syndrome (MPS) is a commonly encountered condition frequently associated with the muscles of mastication. It is defined as a regional muscular pain condition characterized by myofascial trigger points found in one or more muscles and/ or connective tissues. A trigger point is an exquisitely tender spot in discrete taut band of hardened muscle that produce local and referred pain, among other symptoms. Associated symptoms may include muscle weakness, muscle spasm, stiffness, decreased range of motion and autonomic dysfunction. Trigger point can be active i.e. always tender or latent i.e. tender only when palpated.

Any kind of muscle overuse or direct trauma to the muscle can lead to the development of trigger points. Although muscle damage is not required for the development of trigger point, it may be caused by the disruption of the cell membrane, damage to the sarcoplasmic reticulum with a subsequent release of high amounts of calcium ions, and disruption of cytoskeletal proteins, such as desmin, titin and dystrophin. Muscle overuse leads to ATP depletion which causes oxidative stress resulting in local ischemia and lowered pH with subsequent accumulation of inflammatory mediators at these trigger points.

Various therapeutic modalities have been used to treat myofascial trigger points and myofascial pain syndrome including therapeutic ultrasound, muscle stretching, manipulation, acupuncture, occlusal appliances, botulinum injection, pharmacotherapy and dry needling. Platelet rich plasma (PRP) is a newer therapeutic modality for treatment of trigger points. PRP contains many growth factors important for muscle regeneration and myogenesis. The goal of PRP therapy is to concentrate the main growth factors from native blood and to reintroduce them in the injured tissue. Besides healing, it can also decrease pro-inflammatory and apoptotic cells, reducing inflammation. However, still there is paucity of literature and lack of RCT related to use of PRP in trigger points.

So, the present study has been designed to evaluate the efficacy of Platelet Rich Plasma injection in trigger points in masseter muscle in myofascial pain syndrome patients.

ELIGIBILITY:
INCLUSION CRITERIA

The following patients will be included in the study:

1. Patients diagnosed with myofascial pain within masseter muscle as per RDC/TMD (Ia and Ib)
2. Patient's consent for participation in this study.

EXCLUSION CRITERIA

1. Patients with phobia to needles
2. Patients who have undergone previous treatment for myofascial pain in past 3 months
3. Patients with active infection at the site of injection
4. Patients with history of head and neck fracture in the past 6 months.
5. Patients with healing disorder or systemic disease where healing response is compromised
6. Patients on anticoagulant medication
7. Patients with bleeding and clotting disorder
8. Patients with epilepsy/seizures
9. Pregnancy/ Lactation
10. Patients addicted to alcohol/ drug

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-02-24 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
assessment of pain improvement upto 3 months | 3 months
  using Visual Analog Scale score; (0-10); 0 indicates no pain and 10 indicates worst imaginable pain
Maximal Mouth Opening change from baseline to 3 months | 3 months
  measured by digital vernier callipers

SECONDARY OUTCOMES:
Range of Right and left Lateral excursion movements | 3 months
  measured in mm
Range of Protrusive movement | 3 months
  measured in mm
Need for pain medicine utilization | 3 months
  No. of tablets consumed per week
assessment of Patient satisfaction | 3 months
  by Likert scale
assessment of Sleep pattern | 3 months.
  Visual Analog Scale score (0-10); higher score indicates sleep disturbance

CONTACTS AND LOCATIONS:
Locations (1):
- PGIDS, Rohtak, Haryana, India